CLINICAL TRIAL: NCT01330095
Title: Early Administration of Bifidobacterium Bifidum to Very Low Birth Weight Infants: A Pilot Study
Brief Title: Early Administration of Bifidobacterium to Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Women's Medical University (Other)
Responsible Party: Satoshi Kusuda, Tokyo Women's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1016; UMIN000005245 (Other: University hospital Medical Information Network)
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2008-12

CONDITIONS: Preterm Infants
Keywords: Bifidobacterium bifidum; Very low birth weight infant; Enteral feeding; Growth; amount of enteral feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eearly administration (Active Comparator): Administration of Bifidobacterium within 48h after birth
  Interventions: Dietary Supplement: Administration of Bifidobacterium bifidum
- Late administration (Active Comparator): Administration of Bifidobacterium more than 48h after birth
  Interventions: Dietary Supplement: Administration of Bifidobacterium bifidum

INTERVENTIONS:
Dietary Supplement: Administration of Bifidobacterium bifidum — Administration of Bifidobacterium bifidum to very low birth weight infants
  Other Names: Bifidobacterium bifidum OLB6378

SUMMARY:
To evaluate the effects of early administration of probiotics on acceleration of enteral feeding, and on growth of very low birth weight infants, newborn infants with birth weight less than 1500g are administered Bifidobacterium bifidum twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infant

Exclusion Criteria:

* Presence of major congenital malformations

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
the day at total feeding volume reached 100ml/kg/day | post natal day
  the post natal day at total enteral feeding reached 100ml/kg/day

SECONDARY OUTCOMES:
colonizatin of Bifidobacterium | 4 weeks after birth
  the level of Bifidobacterium in feces from the study infants growth rate of the study infants the positive rate of MRSA colonization among the study infants adverse outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo Women's Medical Unversity, Shinjuku, Tokyo, Japan

REFERENCES:
- [Derived] Yamasaki C, Totsu S, Uchiyama A, Nakanishi H, Masumoto K, Washio Y, Shuri K, Ishida S, Imai K, Kusuda S. Effect of Bifidobacterium administration on very-low-birthweight infants. Pediatr Int. 2012 Oct;54(5):651-6. doi: 10.1111/j.1442-200X.2012.03649.x. Epub 2012 Jul 10. PMID 22507386